CLINICAL TRIAL: NCT05761665
Title: Comparison of Kinesiophobia, Balance, Falling and Walking Speeds of the Cognitively Frail Elderly With Alzheimer's Dementia With the Physically Fragile Elderly.
Brief Title: Comparison of Kinesiophobia, Balance, Falling and Walking Speeds of Elderly's With Physical Frailty With Alzheimer's
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Beyza Nur Celik, Physiotherapist, Kırıkkale University
Other Study IDs: KirikkaleU-FTR-BNC
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Alzheimer Disease; Frail Elderly Syndrome
Keywords: Accidental Falls; Alzheimer Disease; Frail Elderly; Frailty; Kinesiophobia; Postural Balance; Walking Speed
MeSH Terms: conditions — Alzheimer Disease; Frailty; Kinesiophobia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Alzheimer: Kinesiophobia, Balance, Falling,Walking Speed and Fragility Will be Evaluated with Tests.
  Interventions: Other: Evaluation
- Physically Fragile: Kinesiophobia, Balance, Falling,Walking Speed and Fragility Will be Evaluated with Tests.
  Interventions: Other: Evaluation
- Healthy: Kinesiophobia, Balance, Falling,Walking Speed and Fragility Will be Evaluated with Tests.
  Interventions: Other: Evaluation

INTERVENTIONS:
Other: Evaluation — Kinesiophobia=Tampa scale Balance=Berg Balance Scale Falling=The Fall Activity Scale( Tinetti) Walking speed=Timed Get Up and Walk Test ,Two-Minute Walking Test Fragility=Frail Fragility Questionnaire, Clinical Fragility Scale

SUMMARY:
In this study, Kinesiophobia, Balance, Falling, Walking Speeds of Elderly People with Cognitive Frailty with Alzheimer's Dementia, Elderly with Physical Frailty and Healthy Elderly Individuals will be compared.

DETAILED DESCRIPTION:
In this study, Kinesiophobia, Balance, Falling, Walking Speeds of Elderly People with Cognitive Frailty with Alzheimer's Dementia, Elderly with Physical Frailty and Healthy Elderly Individuals will be compared.

For research, 3 Groups will be included, including elderly individuals diagnosed with Alzheimer's Dementia, physically fragile elderly individuals and healthy elderly individuals staying at the Private Dikmen Nursing Home and the private Uluçınar Nursing Home. The research will be conducted with a total of 54 individuals who voluntarily participated in the study from June 2023 to February 2024.

The criteria for participation in the study of elderly individuals diagnosed with 1st group Alzheimer's Dementia are to be over 65 years old, to be able to walk independently and to be diagnosed with early or middle stage Alzheimer's by a doctor.

The criteria for participation in the study of physically frail elderly individuals for 2nd group is to be over 65 years old, to be able to walk independently and appearing fragile or pre-frail according to the Frail Questionnaire.

The criteria for participation in the study of the 3rd group of healthy elderly individuals were to be over 65 years old, not to have any psychiatric, neurological and orthopedic problems, and to be able to walk independently.

As a data collection tool; For the descriptive characteristics of the patients, a form containing demographic information will be used. Timed Up and Go Test, Berg Balance Scale, 2 Minutes Walking Test will be used to evaluate balance and gait. Frail Questionnaire and Clinical Frailty Scale will be used for the evaluation of frailty.

Tampa Scale will be used for kinesiophobia assessment. The Fall Activity Scale (Tinetti) will be used to assess the fear of falling. In addition, the cognitive status of individuals will be evaluated with the Mini Mental State Test and the Montreal Cognitive Assessment Test.

ELIGIBILITY:
Inclusion Criteria:

* being over the age of 65 and being able to walk independently.
* Individuals who have been diagnosed with early or mid-stage Alzheimer's by a physician.
* Appearing fragile or pre-frail according to the Frail Questionnaire.

Exclusion Criteria:

* Who has an obstacle to doing physical activity.
* Those who have undergone an operation in the last 6 months.
* Those who do not agree to participate in the research.
* Those who have been diagnosed with late-stage Alzheimer's dementia.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Private Dikmen Nursing Home and Private Ulucınar Nursing Home
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | 6 months
  It is a scale consisting of 14 tests that measure the ability to maintain balance during different positions, postural changes and movement.The assessment is based on the individual's ability to perform each test independently and/or within a specified time or distance.Grading is made between 0 and 4 points. It is expressed as 0 = unable, 4 = normal performance.
  The highest score is 56.0 to 20 points; indicates that the person is wheelchair dependent and has a 100% risk of falling.Between 21-40 points; It indicates that the person can walk with assistance as there is a risk of falling.between 41-56 points; states that they can ambulate independently with very little risk of falling.
  It was designed to evaluate the risk of falling in geriatrics.
Falls efficacy scale(Tinetti) | 6 months
  Tinettti et al. can be measured, the person's activities of daily living (for example, cleaning the house, getting dressed, doing simple shopping, etc.) 10-item questionnaire to evaluate the efficacy level of elderly individuals by looking at their safety.
  They developed the Tinetti Fall Efficiency Scale.How confident are you that you are doing the following activities without falling, while performing daily life activities in 10 different activities "on a scale of 1 to 10, 1 is very confident and 10 is not confident at all?' he does the questioning.Adding the scores gives a total score of 10 (low fall-related activity) to 100 (high fall-related activity).A total score above 70 indicates that the person has a fear of falling.
Tampa Kinesiophobia Scale | 6 months
  It is a 17-item scale developed to measure the fear of movement/re-injury.The scale includes parameters for injury/re-injury and fear-avoidance in work-related activities.Likert 4 points on the scale rating (1= Strongly disagree, 4= I completely agree) is used.4, 8, 12 and After the reversal of Article 16, a total points are calculated.Person between 17-68 total gets a score. The score that the person received on the scale his high level of kinesiophobia is also high shows.
Timed Get Up and Walk Test | 6 months
  The patient is asked to get up from the chair she is sitting on, walk three meters, turn around and sit down again.At this time, the time is recorded.10 seconds and below; the patient walks independently, the risk of falling is very low.11-19 sec.; The patient walks independently, there is a low to moderate risk of falling.20-29 sec. may need help from time to time, there is a moderate to high risk of falling.Over 30 seconds, assistance is needed from time to time and the risk of falling is high.

CONTACTS AND LOCATIONS:
Overall Officials: Meral SERTEL Doc.Dr, Study Director — Kırıkkale University

IPD SHARING:
Plan to Share IPD: No